CLINICAL TRIAL: NCT00299299
Title: Modelling Internal Hepatic Movement With an External Abdominal Marker Block for Use With a Real Time Position Monitoring System for Respiratory Gating
Brief Title: Modelling Internal Hepatic Movement With an External Abdominal Marker
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Jane Lawrence, Royal Marsden NHS Foundation Trust
Other Study IDs: CCR 2736
Record Dates: First submitted 2006-03-03; First posted 2006-03-06 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Patients With Liver Metastases From Colorectal Cancer

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study tests the feasibility and reproducibility of patient-specific motion models. These will be used for quantification of safe margin reduction. Patient-specific motion models will be built by post-processing 4D MRI data with non-rigid registration. By comparing these models between visits, model reproducibility will be assessed, and the methodology refined.

DETAILED DESCRIPTION:
The study will use a real time position management (RPM) system for respiratory gating. The RPM system senses the respiration motion of the patient by tracking a pair of reflective markers on a lightweight "marker block" constructed of a synthetic material. This block is placed on the patient's abdomen.

During Radiotherapy, the beam is only switched on at pre-determined phases of respiration. The appropriate phase of respiration is determined by the RPM system. This implies a reliable correlation of external block motion to internal hepatic movement. This correlation is not a simple one, and requires "modeling".

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma compatible with primary disease in the colon or rectum
* Aged 18 years or older
* Unequivocal contrast-enhanced CT and/or MRI evidence of malignant single or multiple metastases in the liver, metastases at other sites will not be an exclusion criterion
* WHO performance status 0-2 and life expectancy of at least 12 weeks
* Informed written consent

Exclusion Criteria:

* Pregnancy or breast feeding
* Evidence of ascites
* Patients unable for whatever reason to lie flat
* Patients unable to give fully informed consent
* Age< 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 10 RMH patients aged over 18 years with single or multiple hepatic metastases secondary to colorectal cancer. Metastases at other sites will not be an exclusion criterion. WHO performance status 0, 1 or 2.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Dr Diana Tait, Principal Investigator — Royal Marsden HNHS Foundation Trust
Locations (1):
- Royal Marsden Hospital, Chelsea, United Kingdom